CLINICAL TRIAL: NCT03072238
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial Testing Ipatasertib Plus Abiraterone Plus Prednisone/Prednisolone, Relative to Placebo Plus Abiraterone Plus Prednisone/Prednisolone in Adult Male Patients With Asymptomatic or Mildly Symptomatic, Previously Untreated, Metastatic Castrate-Resistant Prostate Cancer
Brief Title: Ipatasertib Plus Abiraterone Plus Prednisone/Prednisolone, Relative to Placebo Plus Abiraterone Plus Prednisone/Prednisolone in Adult Male Patients With Metastatic Castrate-Resistant Prostate Cancer
Acronym: IPATential150
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CO39303; 2016-004429-17 (EudraCT Number)
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Results first posted 2023-04-10 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Prostate Cancer
Keywords: Metastatic Castrate-Resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ipatasertib; abiraterone; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo + Abiraterone (Active Comparator): Participants received Placebo plus Abiraterone (along with Prednisone/Prednisolone), administered orally in 28-day cycles.
  Interventions: Drug: Abiraterone; Drug: Placebo; Drug: Prednisone/Prednisolone
- Ipatasertib + Abiraterone (Experimental): Participants received Ipatasertib plus Abiraterone (along with Prednisone/Prednisolone), administered orally in 28-day cycles.
  Interventions: Drug: Ipatasertib; Drug: Abiraterone; Drug: Prednisone/Prednisolone

INTERVENTIONS:
Drug: Ipatasertib — Oral tablets, 400 mg, given once daily (QD) beginning on Day 1 of Cycle 1 until disease progression or intolerable toxicity.
  Arms: Ipatasertib + Abiraterone
Drug: Abiraterone — Oral tablets of abiraterone, 1000 mg QD, taken on an empty stomach and swallowed whole with water.
Drug: Placebo — Oral tablets (matched to ipatasertib appearance), given QD beginning on Day 1 of Cycle 1 until disease progression or intolerable toxicity.
  Arms: Placebo + Abiraterone
Drug: Prednisone/Prednisolone — Oral tablets of 5 mg, taken twice daily (BID) until disease progression or intolerable toxicity.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics of ipatasertib plus abiraterone and prednisone/prednisolone compared with placebo plus abiraterone and prednisone/prednisolone in participants with metastatic castrate-resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Collaborative Oncology Group (ECOG) performance status of 0 or 1 at screening
* Adequate hematologic and organ function within 28 days before the first study treatment
* Ability to comply with the study protocol, in the investigator's judgment
* Willingness and ability of participants to use the electronic device to report selected study outcomes; Caregivers and site staff can assist with patient diary input but patient must be able to independently comprehend and answer the questionnaires
* Life expectancy of at least 6 months
* Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm
* For enrollment into the China extension cohort, residence in the People's Republic of China

Disease-specific Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma without neuroendocrine differentiation or small-cell features
* Consent to provide a formalin-fixed paraffin-embedded (FFPE) tissue block (preferred) or a minimum of 15 (20 preferred) freshly cut unstained tumor slides from the most recently collected, available tumor tissue accompanied by an associated pathology report (with tumor content information, Gleason score, and disease staging) for PTEN IHC and NGS testing and for other protocol-mandated secondary and exploratory assessments. If only 12-14 slides are available, the patient may still be eligible for the study, after discussion with and approval by the Medical Monitor. Cytologic or fine-needle aspiration samples are not acceptable. Tumor tissue from bone metastases is not acceptable
* A valid PTEN IHC result (testingcentral laboratory tested with results directly sent to IxRS) (e.g., participants with an "invalid" or "failed" PTEN IHC result are not permitted to enroll)
* Metastatic disease documented prior to randomization by clear evidence of bone lesions on bone scan and/or measurable soft tissue disease by computed tomography (CT) and/or magnetic resonance imaging (MRI) (at least one target lesion) according to RECIST v1.1
* Asymptomatic or mildly symptomatic form of prostate cancer
* Progressive disease before initiating study treatment
* Ongoing androgen deprivation with gonadotropin-releasing hormone (GnRH) analog or bilateral orchiectomy, with serum testosterone <= 50 ng/dL (<= 1.7 nmol/L) within 28 days before randomization

Exclusion Criteria:

* Inability or unwillingness to swallow whole pills
* History of malabsorption syndrome or other condition that would interfere with enteral absorption
* Clinically significant history of liver disease consistent with Child-Pugh Class B or C, including cirrhosis, current alcohol abuse, or current known active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Need of more than 10 mg/day of prednisone or an equivalent dose of other anti-inflammatory corticosteroids as a current systemic corticosteroid therapy to treat a chronic disease (e.g., rheumatic disorder)
* Active infection requiring intravenous (IV) antibiotics within 14 days before Day 1, Cycle 1
* Immunocompromised status because of current known active infection with HIV or because of the use of immunosuppressive therapies for other conditions
* Major surgical procedure or significant traumatic injury within 28 days prior to Day 1, Cycle 1, or anticipation of the need for major surgery during study treatment
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias, such as structural heart disease (e.g., severe left ventricular systolic dysfunction, left ventricular hypertrophy), untreated coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), myocardial infarction or atrial thrombotic events within the past 6 months, severe unstable angina, New York Heart Association Class III and IV heart disease or depressed left ventricular ejection fraction (LVEF; previously documented LVEF < 50% without documentation of recovery), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of sudden unexplained death or long QT syndrome
* History of another malignancy within 5 years prior to randomization, except for either adequately treated non-melanomatous carcinoma of the skin, adequately treated melanoma in situ, adequately treated non-muscle-invasive urothelial carcinoma of the bladder (Tis, Ta, and low grade T1 tumors), or other malignancies where the patient has undergone potentially curative therapy with no evidence of disease and are deemed by the treating physician to have a recurrence rate of <5% at 5 years
* Any other diseases, cardiovascular, pulmonary, or metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the participants at high risk from treatment complications.

Disease-Specific Exclusion Criteria:

* Pathologic findings consistent with small-cell or neuroendocrine carcinoma of the prostate
* Any therapy including chemotherapy (e.g., docetaxel) or biological therapy (e.g., vaccine, immunotherapy) for the treatment of castration-resistant prostate cancer. Previous treatment with flutamide, steroidal anti-androgens, androgens, estrogens, bicalutamide, nilutamide, or 5-α reductase inhibitor is permitted.
* Use of opioid medications for cancer-related pain, including codeine and dextropropoxyphene, currently or any time within 4 weeks of Day 1, Cycle 1
* Prior treatment with abiraterone or other known potent CYP17 inhibitors (e.g., ketoconazole, orteronel) or investigational agents that block androgen synthesis. Previous treatment with itraconazole and fluconazole is permitted.
* Prior treatment with enzalutamide or other potent androgen-receptor blockers, approved or experimental (e.g., ARN-509, ODM-201, or galeterone)
* Prior treatment with flutamide (Eulexin®), steroidal anti-androgens (e.g., cyproterone acetate, chlormadinone acetate), androgens, or estrogens treatment within 4 weeks of Cycle 1, Day 1
* Prior treatment with bicalutamide (Casodex®) or nilutamide (Nilandron®) within 6 weeks of Cycle 1, Day 1
* Prior treatment with 5-alpha reductase inhibitors within 4 weeks of Cycle 1, Day 1
* Prior treatment with systemic radiopharmaceuticals (e.g., radium-223 and strontium-89). Radiopharmaceuticals for the purpose of imaging are permitted. Focal palliative radiation to treat cancer-related pain is permitted provided that the last treatment with radiation is at least 14 days prior to Cycle 1, Day 1.
* Prior treatment with approved or experimental therapeutic agents with known inhibition of the PI3K pathway, including PI3K inhibitors, AKT inhibitors, and mTOR inhibitors
* Administration of an investigational therapeutic agent within 28 days of Cycle 1, Day 1
* Known untreated or active central nervous system (CNS) metastases (progressing or requiring anticonvulsant medications or corticosteroids for symptomatic control); a CT or MRI scan of the brain will be performed at screening if required by the local health authority
* Any chronic therapy or use of food supplements that are strong CYP3A4/5 inducers or inhibitors or sensitive substrates of CYP3A or CYP2D6 with a narrow therapeutic window

Abiraterone-Specific Exclusion Criteria:

* Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 95 mmHg)
* History of pituitary or adrenal dysfunction
* Any ongoing cardiac arrhythmias (including atrial fibrillation) that require medical therapy

Ipatasertib-Specific Exclusion Criteria:

* Type 1 or Type 2 diabetes mellitus requiring insulin at study entry
* History of inflammatory bowel disease (e.g., Crohn disease and ulcerative colitis), active bowel inflammation (e.g., diverticulitis)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1101 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2024-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (176):
- United States (32):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - USC Norris Cancer Center, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - Stanford University, Palo Alto, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Lynn Cancer Institute/Boca Raton Regional Hospital, Boca Raton, Florida
  - Miami Cancer Institute of Baptist Health, Inc., Miami, Florida
  - Northside Hospital, Atlanta, Georgia
  - Illinois Cancer Care, Peoria, Illinois
  - Associates in Oncology/Hematology P.C., Rockville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Institute.., Detroit, Michigan
  - HCA Midwest Division, Kansas City, Missouri
  - Urology Cancer Center & GU Research Network, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada (CCCN) - Central Valley, Las Vegas, Nevada
  - Hackensack Univ Medical Center, Hackensack, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Northwest Cancer Specialists, P.C., Tualatin, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Charleston Oncology, P .A, Charleston, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Texas Oncology - Gulf Coast, The Woodlands, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (5):
  - Macquarie University Hospital, Macquarie University, New South Wales
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Monash Medical Centre, EAST Bentleigh, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Eastern Health, Melbourne, Victoria
- Austria (3):
  - Lkh-Univ. Klinikum Graz, Graz
  - Ordensklinikum Linz Elisabethinen, Linz
  - Landeskrankenhaus Salzburg, Salzburg
- Belgium (3):
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - CHU Sart-Tilman, Liège
- Brazil (4):
  - Hospital Luxemburgo, Belo Horizonte, Minas Gerais
  - Liga Norte Riograndense Contra O Câncer, Natal, Rio Grande do Norte
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Canada (8):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Hamilton Health Sciences - Juravinski Cancer Centre, Hamilton, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Hopital Sacre-Coeur Research Centre, Montreal, Quebec
  - CHU de Québec - Université Laval - Hôtel-Dieu de Québec, Québec
- China (6):
  - Beijing Friendship Hospital Affiliated of Capital University of Medical Science, Beijing
  - Jiangsu Cancer Hospital, Nanjing
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Fudan University Shanghai Cancer Center, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
- Costa Rica (2):
  - ICIMED Instituto de Investigación en Ciencias Médicas, San José
  - Clinica CIMCA, San José
- Denmark (2):
  - Aarhus Universitetshospital, Urologisk Afd. K, Aarhus N
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense
- France (13):
  - ICO Paul Papin, Angers
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - CHD Vendée, La Roche-sur-Yon
  - Hopital Claude Huriez, Lille
  - Institut régional du Cancer Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut de cancerologie du Gard, Nîmes
  - Institut Mutualiste Montsouris, Paris
  - CHU Poitiers, Poitiers
  - Hopital d'Instruction des Armees de Begin, Saint-Mandé
  - Hopital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Greece (4):
  - Alexandras Hospital, Athens
  - IASO General Hospital of Athens, Athens
  - University Hospital of Patras Medical Oncology, Pátrai
  - Papageorgiou General Hospital, Thessaloniki
- Hungary (5):
  - Semmelwies University of Medicine, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Budapesti Uzsoki Utcai Kórház, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - B-A-Z County Hospital, Miskolc
- Ireland (4):
  - Cork University Hospital, Cork
  - Adelaide & Meath Hospital, Dublin, Incorporating the National Children's Hospital, Dublin
  - Mater Misericordiae Uni Hospital, Dublin
  - Mater Private Hospital, Dublin
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Meir Medical Center, Kfar Saba
  - Belinson Medical Center, Division of Oncology, Petah Tikva
  - Chaim Sheba medical center, Oncology division, Ramat Gan
- Italy (11):
  - Istituto Nazionale Tumori Irccs Fondazione G. Pascale, Napoli, Campania
  - I.R.S.T Srl IRCCS, Meldola, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena, Modena, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - A.O. Istituti Ospitalieri - Cremona, Cremona, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - A.O. San Carlo Borromeo, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - Ospedale di Trento-Presidio Ospedaliero Santa Chiara, Trento, Trentino-Alto Adige
  - Ospedale Area Aretina Nord, Arezzo, Tuscany
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
- Japan (19):
  - Nagoya University Hospital, Aichi
  - Hirosaki University Hospital, Aomori
  - National Cancer Center East, Chiba
  - Toho University Sakura Medical Center, Chiba
  - Gunma University Hospital, Gunma
  - National Hospital Organization Hokkaido Cancer Center, Hokkaido
  - Kanazawa University Hospital, Ishikawa
  - Yokohama City University Medical Center, Kanagawa
  - Kitasato University Hospital, Kanagawa
  - Kochi Medical School Hospital, Kochi
  - Kumamoto University Hospital, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Niigata University Medical & Dental Hospital, Niigata
  - Kindai University Hospital, Osaka
  - Nippon Medical School Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Keio University Hospital, Tokyo
  - Kyorin University Hospital, Tokyo
  - Yamaguchi University Hospital, Yamaguchi
- Mexico (4):
  - Hospital Angeles Mocel, Mexico City, Mexico CITY (federal District)
  - Centro Medico Culiacan SA de CV, Culiacán, Sinaloa
  - Medical Care & Research, Mérida, Yucatán
  - Consultorio de Especialidad en Urologia Privado, Durango
- Norway (2):
  - Sykehuset Østfold Kalnes, Grålum
  - Akershus universitetssykehus HF, Lørenskog
- Poland (5):
  - Woj. Wielospec. Centrum Onkologii i Traumatologii, ?ód?
  - SPZOZ Opolskie Centrum Onkologii im. Prof. Tadeusza Koszarawskiego, Opole
  - Narodowy Instytut Onkologii im. M. Sklodowskiej-Curie, Warsaw
  - Szpital Grochowski im. dr med. Rafa?a Masztaka Sp. z o.o., Warsaw
  - Dolno?l?skie Centrum Onkologii, Pulmonologii i Hematologii, Wroclaw
- Portugal (3):
  - HUC, Coimbra
  - Hospital de Santa Maria, Lisbon
  - IPO do Porto, Porto
- Russia (4):
  - Altai Regional Oncological Center, Barnaul, Altayskiy Kray
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Blokhin Cancer Research Center, Moscow, Moscow Oblast
  - Privolzhsk Regional Medical Center, Nizhny Novgorod, Niznij Novgorod
- South Korea (6):
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (14):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Institut Catala d?Oncologia Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Insititut Catala D'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (3):
  - Kaohsiung Medical Uni Chung-Ho Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Chang Gung Memorial Hospital-LinKou, Taoyuan District
- Thailand (4):
  - Chulalongkorn Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Faculty of Med. Siriraj Hosp., Bangkok
  - Maharaj Nakorn Chiangmai Hospital, Chiang Mai
- United Kingdom (6):
  - Royal Blackburn Hospital, Blackburn
  - Leicester Royal Infirmary, Leicester
  - The Christie NHS Foundation Trust, Manchester
  - Mount Vernon & Watford Trust Hospital, Northwood
  - Royal Marsden Hospital, Sutton
  - Royal Wolverhampton hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Matsubara N, de Bono J, Sweeney C, Chi KN, Olmos D, Sandhu S, Massard C, Garcia J, Chen G, Harris A, Schenkel F, Sane R, Hinton H, Bracarda S, Sternberg CN. Safety Profile of Ipatasertib Plus Abiraterone vs Placebo Plus Abiraterone in Metastatic Castration-resistant Prostate Cancer. Clin Genitourin Cancer. 2023 Apr;21(2):230-237.e1. doi: 10.1016/j.clgc.2023.01.001. Epub 2023 Jan 7. PMID 36697317
- [Derived] Kotani N, Wilkins JJ, Wade JR, Dang S, Sutaria DS, Yoshida K, Sundrani S, Ding H, Garcia J, Hinton H, Sane R, Chanu P. Characterization of exposure-response relationships of ipatasertib in patients with metastatic castration-resistant prostate cancer in the IPATential150 study. Cancer Chemother Pharmacol. 2022 Dec;90(6):511-521. doi: 10.1007/s00280-022-04488-2. Epub 2022 Oct 28. PMID 36305957
- [Derived] Sweeney C, Bracarda S, Sternberg CN, Chi KN, Olmos D, Sandhu S, Massard C, Matsubara N, Alekseev B, Parnis F, Atduev V, Buchschacher GL Jr, Gafanov R, Corrales L, Borre M, Stroyakovskiy D, Alves GV, Bournakis E, Puente J, Harle-Yge ML, Gallo J, Chen G, Hanover J, Wongchenko MJ, Garcia J, de Bono JS. Ipatasertib plus abiraterone and prednisolone in metastatic castration-resistant prostate cancer (IPATential150): a multicentre, randomised, double-blind, phase 3 trial. Lancet. 2021 Jul 10;398(10295):131-142. doi: 10.1016/S0140-6736(21)00580-8. PMID 34246347

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1101 male participants with metastatic castrate-resistant prostate cancer (mCRPC) took part in the study at 181 investigative sites across 26 countries from June 30, 2017 to April 24, 2024.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to one of the two following treatment arms: abiraterone plus prednisone/prednisolone plus ipatasertib (Ipat + Abi) and abiraterone plus prednisone/prednisolone plus placebo (Pbo + Abi). 3 participants in the Pbo+Abi arm and 1 participant in the Ipat +Abi arm did not receive any treatment. 5 participants randomized to the placebo arm took at least one dose of ipatasertib and hence were included in the Ipat + Abi arm for safety analysis.
Groups:
- Pbo + Abi: Participants received matching placebo along with abiraterone 1000 milligrams (mg), once a day (QD) and prednisone/prednisolone, 5 mg, twice a day (BID) administered orally in each 28 day treatment cycle until disease progression, intolerable toxicity, elective withdrawal from the study, or study completion or termination.
- Ipat + Abi: Participants received ipatasertib, 400 mg, QD along with abiraterone, 1000 mg, QD and prednisone/prednisolone, 5 mg, BID administered orally in each 28 day treatment cycle until disease progression, intolerable toxicity, elective withdrawal from the study, or study completion or termination.
Period: Overall Study
Arm/Group | Pbo + Abi | Ipat + Abi
Started | 554 | 547
Safety Evaluable (SE) Population (SE population included all participants who received any amount of the study treatment. 5 participants randomized to the placebo arm took at least one dose of ipatasertib and hence were included in the Ipat + Abi arm for safety analysis.) | 546 | 551
Completed | 0 | 0
Not Completed | 554 | 547
Not completed — Withdrawal by Subject | 44 | 64
Not completed — Lost to Follow-up | 14 | 5
Not completed — Physician Decision | 4 | 6
Not completed — Death | 351 | 318
Not completed — Progressive Disease | 3 | 4
Not completed — Reason Not Specified | 138 | 150

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all randomized participants, whether or not the participants received the assigned treatment.
Groups:
- Pbo + Abi: Participants received matching placebo along with abiraterone 1000 mg, QD and prednisone/prednisolone, 5 mg, BID administered orally in each 28 day treatment cycle until disease progression, intolerable toxicity, elective withdrawal from the study, or study completion or termination.
- Total: Total of all reporting groups
Arm/Group | Pbo + Abi | Ipat + Abi | Total
Number analyzed (Participants) | 554 | 547 | 1101
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (8.2) | 69.4 (8.0) | 69.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 554 | 547 | 1101
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 65 | 66 | 131
    Not Hispanic or Latino | 469 | 452 | 921
    Not Stated | 13 | 14 | 27
    Unknown | 7 | 15 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    American Indian or Alaska Native | 16 | 15 | 31
    Asian | 109 | 110 | 219
    Black or African American | 9 | 10 | 19
    Native Hawaiian or other Pacific Islander | 1 | 1 | 2
    White | 386 | 376 | 762
    Unknown | 33 | 35 | 68

OUTCOME MEASURES:

1. Primary Outcome: Investigator-assessed Radiographic Progression-free Survival (rPFS), Per Prostate Cancer Working Group 3 (PCWG3) Criteria in Phosphatase and Tensin Homolog (PTEN) Loss Population
Description: rPFS was defined as time from date of randomization to the first occurrence of documented disease progression (PD), as assessed by the investigator with use of the PCWG3 criteria or death from any cause, whichever occurs first. PD for soft tissue was defined as at least a 20% increase in the sum of diameters (SOD) of target lesions, taking as reference the smallest sum on study, including baseline, and an absolute increase of at least 5 millimeters (mm) in the SOD of target lesions; progression of non-target lesions; the appearance of one or more new lesions according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) criteria. PD for bone lesions was defined as 2 or more new lesions compared to baseline followed by a confirmatory bone scan at least 6 weeks later according to the PCWG3 criteria. The Kaplan-Meier (KM) estimate was used to determine the median rPFS.
Time Frame: Up to approximately 32 months
Population: PTEN loss population included all randomized participants with PTEN loss tumors by immunohistochemistry (IHC), regardless of whether or not the participant received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 261 | 260
months | 16.5 [13.9 to 17.0] | 18.5 [16.3 to 22.1]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.0335, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.61 to 0.98]

2. Primary Outcome: Investigator-assessed rPFS, Per PCWG3 Criteria in ITT Population
Description: rPFS was defined as time from date of randomization to the first occurrence of documented PD, as assessed by the investigator with use of the PCWG3 criteria or death from any cause, whichever occurs first. PD for soft tissue was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on study, including baseline, and an absolute increase of at least 5 mm in the SOD of target lesions; progression of non-target lesions; the appearance of one or more new lesions according to RECIST v1.1 criteria. PD for bone lesions was defined as 2 or more new lesions compared to baseline followed by a confirmatory bone scan at least 6 weeks later according to the PCWG3 criteria. The KM estimate was used to determine the median rPFS.
Time Frame: Up to approximately 32 months
Population: ITT population included all randomized participants, whether or not the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 554 | 547
months | 16.6 [15.6 to 19.1] | 19.2 [16.5 to 22.3]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.0431, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.71 to 0.99]

3. Secondary Outcome: Overall Survival (OS) in PTEN-loss Population
Description: OS was defined as the time from randomization to death due to any cause. KM estimates were used to determine the median OS.
Time Frame: Up to approximately 6.5 years
Population: PTEN loss population included all randomized participants with PTEN loss tumors by IHC, regardless of whether or not the participant received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 261 | 260
months | 35.8 [30.8 to 39.6] | 36.8 [31.4 to 42.1]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.5698, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.76 to 1.17]

4. Secondary Outcome: OS in ITT Population
Description: as for outcome 3
Time Frame: Up to approximately 6.5 years
Population: ITT population included all randomized participants, whether or not the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 554 | 547
months | 36.5 [33.9 to 39.4] | 39.4 [36.5 to 42.9]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.2515, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.79 to 1.07]

5. Secondary Outcome: Time to Pain Progression in PTEN-loss Population
Description: Time to pain progression was defined as the time from randomization to the first occurrence of confirmed clinically meaningful cancer-related pain progression event. Cancer-related pain progression refers to pain onset for participants who were asymptomatic at baseline or pain worsening for those who were mildly symptomatic at baseline. Pain severity was graded on a 10-point numeric rating scale [NRS], with 0=no pain and 10=severe pain. Pain severity progression was defined as a ≥ 2-point absolute increase from baseline. KM estimates were used to determine the median time to pain progression.
Time Frame: Up to approximately 5.5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 261 | 260
months | 17.6 [14.6 to 27.7] | 25.8 [17.5 to 43.3]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.6010, Log Rank; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.58 to 1.01]

6. Secondary Outcome: Time to Pain Progression in ITT Population
Description: Time to pain progression was defined as the time from randomization to the first occurrence of confirmed clinically meaningful cancer-related pain progression event. Cancer-related pain progression refers to pain onset for participants who were asymptomatic at baseline or pain worsening for those who were mildly symptomatic at baseline. Pain severity was graded on a 10-point NRS, with 0=no pain and 10=severe pain. Pain severity progression was defined as a ≥ 2-point absolute increase from baseline. KM estimates were used to determine the median time to pain progression.
Time Frame: Up to approximately 5.5 years
Population: ITT population included all randomized participants, whether or not the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 554 | 547
months | 21.9 [17.5 to 27.7] | 25.9 [20.2 to 40.7]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.1723, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.72 to 1.06]

7. Secondary Outcome: Time to Initiation of Cytotoxic Chemotherapy for Prostate Cancer (PC) in PTEN-loss Population
Description: Time to initiation of cytotoxic chemotherapy was defined as the time interval from the date of randomization to the date of initiation of cytotoxic chemotherapy (use of antineoplastic agents: docetaxel, cabazitaxel, mitoxantrone, estramustine, cisplatin, carboplatin, cyclophosphamide, doxorubicin, mitomycin, irinotecan, 5-fluorouracil, gemcitabine, or etoposide) for PC. KM estimates were used to determine the median time to initiation of cytotoxic chemotherapy.
Time Frame: Up to approximately 5.5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 261 | 260
months | 33.6 [26.3 to 38.8] | 36.3 [30.5 to 58.6]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.1566, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.65 to 1.07]

8. Secondary Outcome: Time to Initiation of Cytotoxic Chemotherapy for PC in ITT Population
Description: as for outcome 7
Time Frame: Up to approximately 5.5 years
Population: ITT population included all randomized participants, whether or not the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 554 | 547
months | 35.5 [30.9 to 40.3] | 40.4 [34.7 to NA] — The upper limit of 95% confidence interval (CI) was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.0419, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.69 to 0.99]

9. Secondary Outcome: Time to Function Deterioration Per European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) Physical Function (PF) Scale and Role Function (RF) Scale in PTEN-loss Population
Description: Time to function deterioration=time from date of randomization to date of 10-point or more score decrease on either EORTC QLQ-C30 5-item PF/2-item RF scale scores, held for two consecutive assessments or death within 28 days, whichever occurs first. EORTC QLQ-C30 consists of 30 questions that assess 5 aspects of participant functioning (physical,emotional,role,cognitive&social), 3 symptom scales (fatigue,nausea&vomiting,pain), global health/quality of life (GHS/QoL)&6 single items (dyspnea,insomnia,appetite loss,constipation,diarrhea&financial difficulties). PF scale has 5 questions about participants physical functioning&daily activities. RF scale has 2 questions about work/daily activities&hobbies/leisurely activities. PF&RF are scored on a 4-point scale (1=Not at All to 4=Very Much). Obtained scores are linearly transformed to score range of 0-100, where higher scores indicate a higher response level (better PF)&better functioning/support.
Time Frame: Up to approximately 5.5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 261 | 260
months | 15.7 [12.1 to 21.2] | 12.5 [9.3 to 16.3]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.3198, Log Rank; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.89 to 1.45]

10. Secondary Outcome: Time to Function Deterioration Per EORTC QLQ-C30 PF Scale and RF Scale in ITT Population
Description: Time to function deterioration=time from date of randomization to date of 10-point or more score decrease on either EORTC QLQ-C30 5-item PF/2-item RF scale scores, held for two consecutive assessments or death within 28 days, whichever occurs first. EORTC QLQ-C30 consists of 30 questions that assess 5 aspects of participant functioning (physical,emotional,role,cognitive & social), 3 symptom scales (fatigue,nausea&vomiting,pain), GHS/QoL & 6 single items (dyspnea,insomnia,appetite loss,constipation,diarrhea & financial difficulties). PF scale has 5 questions about participants physical functioning & daily activities. RF scale has 2 questions about work/daily activities & hobbies/leisurely activities. PF&RF are scored on a 4-point scale (1=Not at All to 4=Very Much). Obtained scores are linearly transformed to score range of 0-100, where higher scores indicate a higher response level (better PF) & better functioning/support.
Time Frame: Up to approximately 5.5 years
Population: ITT population included all randomized participants, whether or not the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 554 | 547
months | 14.8 [12.0 to 18.2] | 9.2 [7.4 to 11.1]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.0071, Log Rank; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [1.06 to 1.47]

11. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression, Per the PCWG3 Criteria in PTEN-loss Population
Description: Time to PSA progression was defined as the time from the date of randomization to the first occurrence of PSA progression, per the PCWG3 criteria. PSA progression was defined as a PSA increase that was ≥ 25% and ≥ 2 nanograms per milliliters (ng/mL) above the baseline or the nadir, which was confirmed by a second value ≥ 3 weeks later. KM estimate was used to determine the median time to PSA.
Time Frame: Up to approximately 5.5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 261 | 260
months | 7.6 [6.5 to 9.3] | 12.6 [10.2 to 15.3]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.0045, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.59 to 0.91]

12. Secondary Outcome: Time to PSA Progression, Per the PCWG3 Criteria in ITT Population
Description: Time to PSA progression was defined as the time from the date of randomization to the first occurrence of PSA progression, per the PCWG3 criteria. PSA progression was defined as a PSA increase that was ≥ 25% and ≥ 2 ng/mL above the baseline or the nadir, which was confirmed by a second value ≥ 3 weeks later. KM estimate was used to determine the median time to PSA.
Time Frame: Up to approximately 5.5 years
Population: ITT population included all randomized participants, whether or not the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 554 | 547
months | 8.3 [7.4 to 9.3] | 12.6 [10.3 to 14.8]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.61 to 0.83]

13. Secondary Outcome: Time to First Opioid Use in PTEN-loss Population
Description: Time to first opioid use was defined as the time interval from the date of randomization to the date of an initiation of opioid analgesic use for cancer-related pain, and consumption reported on at least 7 consecutive days. KM estimate was used to determine the median time to first opioid use.
Time Frame: Up to approximately 5.5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 261 | 260
months | NA [14.1 to NA] — The median and upper limit of 95% CI were not estimable due to insufficient number of participants with events. | NA [21.5 to NA] — The median and upper limit of 95% CI were not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.1359, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.57 to 1.08]

14. Secondary Outcome: Time to First Opioid Use in ITT Population
Description: as for outcome 13
Time Frame: Up to approximately 5.5 years
Population: ITT population included all randomized participants, whether or not the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 554 | 547
months | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of participants with events. | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.1398, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.68 to 1.06]

15. Secondary Outcome: Time to Symptomatic Skeletal Event (SSE) in PTEN-loss Population
Description: Time to SSE was defined as the time from randomization to the first occurrence of an SSE. A SSE was defined using one of the following: use of external-beam radiotherapy to relieve skeletal symptoms (including initiation of radium-223 to treat symptoms of bone metastases); occurrence of a new symptomatic pathological bone fracture (vertebral or non-vertebral); clinically apparent occurrence of spinal cord compression, or a tumor-related orthopedic surgical intervention. KM estimates were used to determine the median time to SSE.
Time Frame: Up to approximately 5.5 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 261 | 260
months | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of participants with events. | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.8239, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.61 to 1.48]

16. Secondary Outcome: Time to SSE in ITT Population
Description: as for outcome 15
Time Frame: Up to approximately 5.5 years
Population: ITT population included all randomized participants, whether or not the participants received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 554 | 547
months | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of participants with events. | NA [NA to NA] — The median and 95% CI were not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.6018, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.66 to 1.27]

17. Secondary Outcome: Objective Response Rate (ORR) Per RECIST V1.1 and PCWG3 Criteria in Participants With Measurable Disease in PTEN-loss Population
Description: ORR was defined as the percentage of participants who had an objective response (OR) with measurable disease at baseline. An OR was defined as a complete response (CR) or partial response (PR) on two consecutive occasions ≥ 4 weeks apart, as determined by the investigator using RECIST v1.1 and PCWG3 criteria in participants with measurable disease at baseline. CR was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have a reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. An estimate of ORR was calculated for each treatment arm, and its 95% CI was calculated using the Clopper-Pearson method. Percentages have been rounded off.
Time Frame: Up to approximately 5.5 years
Population: PTEN loss population included all randomized participants with PTEN loss tumors by IHC, regardless of whether or not the participant received the assigned treatment. Overall number analyzed is the number of participants with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 96 | 99
percentage of participants | 42.7 [32.66 to 53.22] | 63.6 [53.36 to 73.07]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.0030, Cochran-Mantel-Haenszel; Difference in Overall Response Rate = 20.93, 95% CI 2-sided [6.20 to 35.65]

18. Secondary Outcome: ORR Per RECIST V1.1 and PCWG3 Criteria in Participants With Measurable Disease in ITT Population
Description: ORR was defined as the percentage of participants who had an OR with measurable disease at baseline. An OR was defined as a CR or PR on two consecutive occasions ≥ 4 weeks apart, as determined by the investigator using RECIST v1.1 and PCWG3 criteria in participants with measurable disease at baseline. CR was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have a reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. An estimate of ORR was calculated for each treatment arm, and its 95% CI was calculated using the Clopper-Pearson method. Percentage have been rounded off.
Time Frame: Up to approximately 5.5 years
Population: ITT population included all randomized participants, whether or not the participants received the assigned treatment. Overall number analyzed is the number of participants with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 225 | 201
percentage of participants | 46.2 [39.57 to 52.97] | 62.7 [55.60 to 69.39]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel; Difference in Overall Response Rate = 16.46, 95% CI 2-sided [6.66 to 26.27]

19. Secondary Outcome: Duration of Confirmed Response (DOCR) in PTEN-loss Population
Description: DOCR was defined as the time from the first documented OR (CR or PR) to documented PD as determined by the investigator using RECIST v1.1 and PCWG3 criteria, or death from any cause, whichever occurred first. CR was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on study, including baseline, and an absolute increase of at least 5 mm in the SOD of target lesions; progression of non-target lesions; the appearance of one or more new lesions. DOR was estimated using the KM methodology.
Time Frame: Up to approximately 5.5 years
Population: PTEN loss population included all randomized participants with PTEN loss tumors by IHC, regardless of whether or not the participant received the assigned treatment. Overall number analyzed is the number of participants with objective response i.e. responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 41 | 63
months | 14.4 [12.1 to 18.5] | 19.6 [15.3 to 24.4]

20. Secondary Outcome: DOCR in ITT Population
Description: DOCR was defined as the time from the first documented OR (CR or PR) to documented PD as determined by the investigator using RECIST v1.1 and PCWG3 criteria, or death from any cause, whichever occured first. CR was defined as disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on study, including baseline, and an absolute increase of at least 5 mm in the SOD of target lesions; progression of non-target lesions; the appearance of one or more new lesions. DOR was estimated using the KM methodology.
Time Frame: Up to approximately 5.5 years
Population: ITT population included all randomized participants, whether or not the participants received the assigned treatment. Overall number analyzed is the number of participants with objective response i.e. responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 104 | 126
months | 16.3 [13.4 to 20.2] | 18.2 [14.4 to 22.1]

21. Secondary Outcome: PSA Response Rate in PTEN-loss Population
Description: PSA response rate was defined as the percentage of participants achieving a PSA decline ≥ 50% from baseline. Participants without a post-baseline PSA assessment were considered to be non-responders. Percentages have been rounded off.
Time Frame: Up to approximately 5.5 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 261 | 260
percentage of participants | 71.6 [65.76 to 77.03] | 83.5 [78.38 to 87.77]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.0012, Cochran-Mantel-Haenszel; Difference in Overall Response Rate = 11.81, 95% CI 2-sided [4.34 to 19.29]

22. Secondary Outcome: PSA Response Rate in ITT Population
Description: as for outcome 21
Time Frame: Up to approximately 5.5 years
Population: ITT population included all randomized participants, whether or not the participants received the assigned treatment. Overall number analyzed included participants with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 554 | 546
percentage of participants | 75.5 [71.65 to 78.98] | 81.3 [77.79 to 84.50]
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.0178, Cochran-Mantel-Haenszel; Difference in Overall Response Rate = 5.87, 95% CI 2-sided [0.83 to 10.90]

23. Secondary Outcome: Investigator-assessed rPFS Per PCWG3 Criteria in PTEN-loss Population by Next-generation Sequencing (NGS)
Description: rPFS was defined as time from date of randomization to the first occurrence of documented PD, as assessed by the investigator using the PCWG3 criteria or death from any cause, whichever occurs first. PD for soft tissue was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on study, including baseline, and an absolute increase of at least 5 mm in the SOD of target lesions; progression of non-target lesions; the appearance of one or more new lesions. PD for bone lesions was defined as 2 or more new lesions compared to baseline followed by a confirmatory bone scan at least 6 weeks later.
Time Frame: Up to approximately 32 months
Population: PTEN loss population included all randomized participants with PTEN loss tumors by NGS, regardless of whether or not the participant received the assigned treatment. Number analyzed is the number of participants with data available for analyses.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 103 | 105
months | 14.2 [10.9 to 18.7] | 19.1 [13.9 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pbo + Abi vs Ipat + Abi; Test type: Superiority; p = 0.0246, Log Rank; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.45 to 0.95]

24. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study were also considered as AEs. Percentages have been rounded off.
Time Frame: Up to 28 days after last study drug administration (approximately 6.5 years)
Population: SE population included all participants who received any amount of the study treatment. 5 participants randomized to the placebo arm took at least one dose of ipatasertib and hence were included in the Ipat + Abi arm for safety analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 546 | 551
percentage of participants | 96.2 | 99.6

25. Secondary Outcome: Plasma Concentrations of Ipatasertib at Specified Timepoints
Description: Plasma samples for pharmacokinetic characterization was collected at various timepoints in all participants.
Time Frame: 1-3 hours post-dose (Cycle 1, Day 1; Cycle 1 Day 15 and Cycle 3 Day 1) and pre-dose at steady state (Cycle 1 Day 15, Cycle 3 Day 1, Cycle 6 Day 1) (each cycle length= 28 days)
Population: Pharmacokinetic (PK)-evaluable population included all participants who received ipatasertib treatment with evaluable PK samples. Number analyzed per timepoint are unique number of participants out all the assessed participants with data available for analysis at the specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ipat + Abi
Number analyzed (Participants) | 544
ng/mL
  Cycle 1 Day 1 Post-dose: number analyzed (Participants) | 499
  Cycle 1 Day 1 Post-dose | 212 (158)
  Cycle 1 Day 15 Pre-dose: number analyzed (Participants) | 467
  Cycle 1 Day 15 Pre-dose | 46.8 (160)
  Cycle 1 Day 15 Post-dose: number analyzed (Participants) | 413
  Cycle 1 Day 15 Post-dose | 247 (138)
  Cycle 3 Day 1 Pre-dose: number analyzed (Participants) | 407
  Cycle 3 Day 1 Pre-dose | 35.4 (256)
  Cycle 3 Day 1 Post-dose: number analyzed (Participants) | 403
  Cycle 3 Day 1 Post-dose | 207 (156)
  Cycle 6 Day 1 Pre-dose: number analyzed (Participants) | 372
  Cycle 6 Day 1 Pre-dose | 46.1 (134)

26. Secondary Outcome: Plasma Concentrations of Abiraterone at Specified Timepoints
Description: Plasma samples for pharmacokinetic characterization was collected at various timepoints in all participants.
Time Frame: Pre-dose at steady state in Cycle 1, Day 15 and Cycle 3 Day 1 (each cycle length= 28 days)
Population: PK-evaluable population included all participants who received abiraterone treatment with evaluable PK samples. Overall number analyzed is the number of participants with data available for analysis. Number analyzed are unique number of participants out of all the assessed participants with data available at the specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pbo + Abi | Ipat + Abi
Number analyzed (Participants) | 537 | 520
ng/mL
  Cycle 1 Day 15: number analyzed (Participants) | 508 | 470
  Cycle 1 Day 15 | 11.2 (124) | 9.40 (159)
  Cycle 3 Day 1: number analyzed (Participants) | 492 | 415
  Cycle 3 Day 1 | 10.4 (120) | 9.55 (159)

ADVERSE EVENTS:
Time Frame: Up to approximately 6.5 years
Description: SE Population included all participants who received any amount of the study treatment. 5 participants randomized to the placebo arm took at least one dose of ipatasertib and hence were included in the Ipat + Abi arm for safety analysis.
Arm/Group | Pbo + Abi | Ipat + Abi
All-Cause Mortality (participants affected / at risk) | 358/546 | 331/551
Serious Adverse Events (participants affected / at risk) | 158/546 | 252/551
Other Adverse Events (participants affected / at risk) | 496/546 | 541/551
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pbo + Abi (N=546) | Ipat + Abi (N=551)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 7 (7)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 7 (7) | 3 (3)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 4 (4)
Cardiac failure (Cardiac disorders) | 1 (1) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (4) | 7 (7)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 14 (14)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 2 (2)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ischaemic enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 1 (1) | 1 (1)
Death (General disorders) | 3 (3) | 4 (4)
Fatigue (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 2 (2)
Hernia (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 4 (4)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 2 (2)
Haemobilia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2) | 2 (2)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Bullous erysipelas (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 5 (5)
Cellulitis (Infections and infestations) | 3 (3) | 3 (3)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Opportunistic infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 10 (10) | 16 (17)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (3) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 2 (3)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 6 (6) | 6 (6)
Septic shock (Infections and infestations) | 0 (0) | 5 (5)
Skin infection (Infections and infestations) | 0 (0) | 2 (3)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 6 (6) | 12 (15)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (6) | 2 (2)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypobarism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumonitis chemical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 5 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 12 (13)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 25 (26)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 2 (2)
Spinal cord compression (Nervous system disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 2 (3) | 2 (2)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 5 (5)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 6 (7) | 11 (13)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 3 (3)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (3)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 3 (3)
Urinary tract obstruction (Renal and urinary disorders) | 3 (3) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 15 (17)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Artery dissection (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Superior mesenteric artery dissection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Bacterial abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 6 (6)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 1 (1)
Prostate infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Sacral pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Benign neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary fistula (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pbo + Abi (N=546) | Ipat + Abi (N=551)
Anaemia (Blood and lymphatic system disorders) | 75 (107) | 127 (192)
Abdominal pain (Gastrointestinal disorders) | 22 (24) | 32 (38)
Constipation (Gastrointestinal disorders) | 95 (111) | 55 (60)
Diarrhoea (Gastrointestinal disorders) | 137 (193) | 441 (969)
Dyspepsia (Gastrointestinal disorders) | 27 (33) | 37 (40)
Nausea (Gastrointestinal disorders) | 65 (76) | 159 (214)
Vomiting (Gastrointestinal disorders) | 57 (75) | 98 (152)
Asthenia (General disorders) | 78 (99) | 103 (148)
Fatigue (General disorders) | 111 (141) | 129 (148)
Oedema peripheral (General disorders) | 56 (73) | 89 (105)
Pyrexia (General disorders) | 23 (26) | 38 (45)
Nasopharyngitis (Infections and infestations) | 52 (72) | 48 (68)
Upper respiratory tract infection (Infections and infestations) | 50 (60) | 39 (52)
Urinary tract infection (Infections and infestations) | 46 (61) | 54 (87)
Fall (Injury, poisoning and procedural complications) | 53 (72) | 42 (58)
Alanine aminotransferase increased (Investigations) | 56 (67) | 110 (129)
Aspartate aminotransferase increased (Investigations) | 58 (71) | 94 (101)
Blood creatinine increased (Investigations) | 27 (35) | 41 (56)
Weight decreased (Investigations) | 23 (27) | 78 (94)
Decreased appetite (Metabolism and nutrition disorders) | 62 (78) | 107 (128)
Hyperglycaemia (Metabolism and nutrition disorders) | 95 (155) | 220 (366)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 28 (36) | 36 (43)
Hypokalaemia (Metabolism and nutrition disorders) | 44 (69) | 48 (70)
Arthralgia (Musculoskeletal and connective tissue disorders) | 119 (155) | 102 (139)
Back pain (Musculoskeletal and connective tissue disorders) | 127 (164) | 105 (135)
Bone pain (Musculoskeletal and connective tissue disorders) | 37 (52) | 47 (52)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 56 (68) | 45 (54)
Dizziness (Nervous system disorders) | 35 (46) | 41 (47)
Headache (Nervous system disorders) | 48 (62) | 58 (68)
Insomnia (Psychiatric disorders) | 44 (50) | 29 (31)
Haematuria (Renal and urinary disorders) | 33 (41) | 35 (50)
Cough (Respiratory, thoracic and mediastinal disorders) | 50 (55) | 47 (52)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 (31) | 36 (37)
Pruritus (Skin and subcutaneous tissue disorders) | 16 (18) | 48 (66)
Rash (Skin and subcutaneous tissue disorders) | 48 (53) | 150 (193)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (9) | 48 (67)
Hot flush (Vascular disorders) | 38 (42) | 28 (31)
Hypertension (Vascular disorders) | 94 (125) | 86 (102)
Blood alkaline phosphatase increased (Investigations) | 28 (32) | 27 (29)
Blood cholesterol increased (Investigations) | 12 (12) | 28 (37)
Glycosylated haemoglobin increased (Investigations) | 7 (7) | 30 (32)
Lipase increased (Investigations) | 27 (44) | 30 (48)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 15 (20) | 33 (36)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 32 (34) | 21 (28)
Dysuria (Renal and urinary disorders) | 20 (23) | 30 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT03072238/Prot_002.pdf
  • Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT03072238/SAP_001.pdf